CLINICAL TRIAL: NCT00848939
Title: An Evaluation of the Pharmacokinetics and Safety of Fixed and Escalating Doses of Oral Treprostinil Diethanolamine (UT-15C) Sustained Release Tablets in Patients With Systemic Sclerosis
Brief Title: Pharmacokinetics of Oral Treprostinil in Patients With Systemic Sclerosis
Acronym: DISTOL-PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDE-DU-101
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis; scleroderma; pharmacokinetics; treprostinil diethanolamine
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treprostinil diethanolamine (Experimental)
  Interventions: Drug: treprostinil diethanolamine

INTERVENTIONS:
Drug: treprostinil diethanolamine — Cohort 1: Single 1 mg treprostinil diethanolamine sustained release tablet dose
Drug: treprostinil diethanolamine — Cohort 2: treprostinil diethanolamine sustained release doses will be escalated up to a target dose of 4 mg BID

SUMMARY:
This study will assess the pharmacokinetic and safety profile of treprostinil following fixed and escalating doses of treprostinil diethanolamine SR tablets. Open-label, two-part study assessing the pharmacokinetics, safety, and tolerability of oral treprostinil diethanolamine SR. Cohort 1: single 1 mg treprostinil diethanolamine SR dose. Cohort 2: escalating doses of treprostinil diethanolamine SR up to a target dose of 4 mg BID.

ELIGIBILITY:
Inclusion Criteria:

* Subject gives voluntary written informed consent to participate in the study.
* Subject has been diagnosed with systemic sclerosis (SSc) as defined by American College of Rheumatology (ACR) criteria.
* Males and females age greater than 18 years at time of Screening.
* Presence of active digital ulcer OR history of digital ulcer occurring within past 6 months at time of Screening and poorly controlled Raynaud's phenomenon (as documented by patient report of 6-10 episodes per week).
* Females of childbearing potential must be willing to use two forms of medically acceptable contraception (at least one barrier method) and have a negative pregnancy test at Screening, confirmed at Baseline if separate visits. Women who are surgically sterile or have been post-menopausal for at least 2 years are not considered to be of child-bearing potential.
* Subject agrees to abstain from consuming grapefruit containing food or beverages for 3 days prior to Baseline and until discharge from the study.
* Subject is able to communicate effectively with study personnel and be considered reliable, willing and cooperative in terms of compliance with the protocol requirements.

Exclusion Criteria:

* Has diagnosis of pulmonary arterial hypertension and receiving approved or investigational therapies for PAH, including endothelin receptor antagonists, phosphodiesterase inhibitors, or prostacyclin analogues.
* Body weight less than 40 kg at time of Screening, confirmed at Baseline.
* The subject has a history of postural hypotension, unexplained syncope, a blood pressure that is less than 85 mmHg systolic or 50 mmHg diastolic at Screening or Baseline.
* Hemoglobin concentration less than 75% of the lower limit of the normal range at time of Screening.
* AST and/or ALT concentrations greater than 3 times upper limit of normal (ULN) at time of Screening.
* Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C.
* Intractable diarrhea, severe malabsorption, defined as greater than 15% unintentional loss of body weight in the last 6 months prior to Screening, or any severe organ failure (e.g., lung, kidney) or any life-threatening condition.
* Pregnancy or breast-feeding.
* Overlap with another connective tissue disease that could affect rest pain and hand function (e.g. diabetes mellitus, rheumatoid arthritis).
* Sympathectomy of the upper limb performed within 12 months of Baseline.
* Receipt of parenteral prostanoid treatment (epoprostenol, treprostinil sodium, or other prostacyclin analog) within the previous 3 months for conditions including PAH, rest pain and / or digital ulcers.
* Treatment with gemfibrozil, glitazones, or cyclophosphamide within 1 week prior to Baseline.
* Treatment with rifampin within 4 weeks prior to Baseline.
* Local injection of botulinum toxin in an affected finger within 1 month prior to Baseline.
* Received systemic antibiotics to treat infection of digital ulcers within 2 weeks prior to Baseline.
* Treatment with phosphodiesterase inhibitors such as sildenafil, except for intermittent treatment of male erectile dysfunction.
* Received an investigational product within 1 month preceding Screening.
* Known hypersensitivity to oral treprostinil or any of the excipients.
* Cigarette smoking at any level within the past 6 months prior to Screening.
* Any condition that could prevent compliance with the protocol or adherence to therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Cohort 1: treprostinil pharmacokinetics in patients with systemic sclerosis following single oral administration of a 1 mg treprostinil diethanolamine SR dose. | pre-24hrs post dose
Cohort 2: treprostinil pharmacokinetics at dose levels of 2 mg BID and 4 mg BID, respectively, in patients with systemic sclerosis following repeated oral administration of treprostinil diethanolamine SR tablets | 0-12 hrs post-dose
adverse event monitoring | Cohort 1:Day 0 to Day 2; Cohort 2: Day 0 to Day 47

SECONDARY OUTCOMES:
clinical laboratories | Cohort 1: Day 0 and Day 2; Cohort 2: Day 0 and Day 47
Cohort 2: Raynauds Phenomenon Visual Analoge Scale | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kristan Rollins, PharmD, Study Director — United Therapeutics
Locations (3):
- United States (3):
  - Johns Hopkins Scleroderma Center, Baltimore, Maryland
  - Boston University School of Medicine Rheumatology Arthritis Center, Boston, Massachusetts
  - University of Michigan Scleroderma Program, Ann Arbor, Michigan

REFERENCES:
- [Derived] Shah AA, Schiopu E, Hummers LK, Wade M, Phillips K, Anderson C, Wise R, Boin F, Seibold JR, Wigley F, Rollins KD. Open label study of escalating doses of oral treprostinil diethanolamine in patients with systemic sclerosis and digital ischemia: pharmacokinetics and correlation with digital perfusion. Arthritis Res Ther. 2013 Apr 18;15(2):R54. doi: 10.1186/ar4216. PMID 23597147